CLINICAL TRIAL: NCT05509699
Title: An Open-Label, Multi-Center Phase II Study of Surufatinib Plus Anti-PD-1/L1 as Maintenance Therapy in Patients With Extensive-Stage Small Cell Lung Cancer
Brief Title: Surufatinib Plus Anti-PD-1/L1 as Maintenance Therapy in Extensive-Stage Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hutchison Medipharma Limited (Industry)
Responsible Party: Sponsor
Organization: Hutchmed (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-012-00CH1
Record Dates: First submitted 2022-08-16; First posted 2022-08-22 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Extensive-Stage Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — surufatinib; Immune Checkpoint Inhibitors

STUDY DESIGN:
Intervention Model Description: The study consists of two parts, i.e., a single-arm Phase IIa study and a randomized (1:1), controlled Phase IIb study.
  Phase IIa:
  It is planned that 20 patients will be enrolled to receive treatment with Surufatinib plus anti-PD-1/L1, the same immune checkpoint inhibitor from patients' first-line therapy .
  Phase IIb:
  It is planned that 40 patients will be enrolled to receive the following treatments:
  Group A: Patients will receive treatment with Surufatinib plus anti-PD-1/L1, the same immune checkpoint inhibitor from patients' first-line therapy.
  Group B: Patients will receive treatment with anti-PD-1/L1, the same immune checkpoint inhibitor from patients' first-line therapy.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Surufatinib in combination with anti-PD-1/L1 therapy (Experimental): Surufatinib 250 mg orally once plus anti-PD-1/L1, Q3W or Q4W, the same immune checkpoint inhibitor from patients' first-line therapy.
  Interventions: Drug: Surufatinib; Drug: Anti-PD-1/L1
- Anti-PD-1/L1 monotherapy (Experimental): Anti-PD-1/L1 therapy, Q3W or Q4W, the same immune checkpoint inhibitor from patients' first-line therapy
  Interventions: Drug: Anti-PD-1/L1

INTERVENTIONS:
Drug: Surufatinib — The recommended dosage is 250 mg orally once daily (QD) within 1 hour after breakfast for continuous administration.
  Arms: Surufatinib in combination with anti-PD-1/L1 therapy
Drug: Anti-PD-1/L1 — Anti-PD-1/L1 therapy, Q3W or Q4W, the same immune checkpoint inhibitor from patients' first-line therapy.
  Other Names: Immune checkpoint inhibitor

SUMMARY:
This is an open-label, multi-center Phase II study designed to evaluate the efficacy and safety of Surufatinib plus anti-PD-1/L1 as maintenance therapy after first-line standard of care in patients with ES-SCLC.

DETAILED DESCRIPTION:
This study consists of two parts, i.e., a single-arm Phase IIa study and a randomized, controlled Phase IIb study. All the enrolled patients will be patients with ES-SCLC who did not have PD (determined as per the RECIST v1.1) after prior platinum-based chemotherapy in combination with an anti-PD-1/L1. Approximately 20 patients are planned to be enrolled in the single-arm Phase IIa study to preliminarily observe the efficacy and safety. Approximately 40 patients are planned to be enrolled in the randomized and controlled Phase IIb study with 20 patients per group.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who sufficiently understand this study and is willing to sign the ICF;
2. Aged from 18 to 75 years (inclusive);
3. Patients with histologically or cytologically confirmed ES-SCLC ;
4. Patients who did not have PD (assessed as per the RECIST v1.1) after prior first-line platinum-based chemotherapy plus an anti-PD-1/L1;
5. Patients with measurable lesions as defined in the RECIST v1.1 ;
6. Life expectancy ≥ 12 weeks;
7. Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 to 1;
8. Adequate organ function:
9. Females of childbearing potential must have a negative serum pregnancy test within 7 days prior to the first dose. Male or female patients of childbearing potential should be willing to use effective contraceptive methods during the study and within 90 days after last dose of the study drug.

Exclusion Criteria:

1. Previous use of anti-vascular endothelial growth factor (VEGF) drugs/anti-vascular endothelial growth factor receptor (VEGFR) agents;
2. Use of systematic anti-tumor therapies other than first-line platinum-based chemotherapy in combination with anti-PD-1/L1 within 4 weeks prior to the first dose;
3. Presence of central nervous system (CNS) metastasis and/or cancerous meningitis (metastases to meninges);
4. Toxicities associated with previous anti-tumor treatment that has not been resolved to CTCAE Grade ≤ 1, except for alopecia and CTCAE Grade ≤ 2 peripheral neurotoxicity;
5. Uncontrollable malignant hydrothorax, ascites or pericardial effusion;
6. Patients with active autoimmune disorder or immunodeficiency or history of autoimmune disorder or immunodeficiency;
7. Patients with evidence or history of obvious bleeding tendency within 2 months prior to the first dose;
8. Clinically significant cardiovascular disorders;
9. Severe infection within 4 weeks prior to the start of study treatment, including but not limited to hospitalization for infection, bacteraemia or severe pneumonia;
10. Patients who are unable to take oral medications, or with previous surgical history or severe gastrointestinal;
11. Pregnant (with a positive pregnancy test) or lactating women within 5 years before screening.
12. Patients with a history of malignant tumors excluding small cell lung cancer (SCLC) within 5 years before screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-09-27 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | About 18 months
  Progression-free survival(PFS) assessed by the investigator as per the Response Evaluation Criteria in Solid Tumors v1.1 (RECIST v1.1)

SECONDARY OUTCOMES:
Overall survival | About 18 months
  Overall survival (OS)
Objective response rate | About 18 months
  Objective response rate (ORR) assessed per RECIST v1.1
Disease control rate | About 18 months
  Disease control rate (DCR) assessed per RECIST v1.1
Duration of response | About 18 months
  Duration of response (DoR) assessed per RECIST v1.1

CONTACTS AND LOCATIONS:
Overall Officials: Yi Hu, Postdoctor, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, China